CLINICAL TRIAL: NCT02190461
Title: Impact of Early Respiratory Rehabilitation in the Exacerbations of Re-admitted Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Impact of Early Respiratory Rehabilitation in the Exacerbations of Re-admitted COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Spanish Society of Pneumology and Thoracic Surgery (Other); Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-EXA-2013-04
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Early Respiratory Rehabilitation; Chronic Obstructive Pulmonary Disease; Re-admitted patients; Open clinical trial; Exacerbations
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Respiratory Rehabilitation (Experimental): Starting the Early Respiratory Rehabilitation programme during the admission and continues it at home immediately after discharge for a period of 3 months.
  Interventions: Procedure: Early Respiratory Rehabilitation Program
- Conventional Respiratory Rehabilitation (Active Comparator): Started a conventional Respiratory Rehabilitation programme at home one month after discharge from hospital and continues for 3 months.
  Interventions: Procedure: Conventional Respiratory Rehabilitation Program

INTERVENTIONS:
Procedure: Early Respiratory Rehabilitation Program
  Arms: Early Respiratory Rehabilitation
Procedure: Conventional Respiratory Rehabilitation Program
  Arms: Conventional Respiratory Rehabilitation

SUMMARY:
Open clinical trial with 1 year follow up comparing the impact of an Early Respiratory Rehabilitation program with the conventional Respiratory Rehabilitation in COPD re-admitted patients. Outcomes will be exacerbations, symptoms, functional capacity and quality of life related to health (HRQOL).

DETAILED DESCRIPTION:
Open clinical trial with 1 year follow up comparing the impact of an Early Respiratory Rehabilitation (ERR) program with the conventional Respiratory Rehabilitation (CRR) in COPD re-admitted patients. Outcomes will be exacerbations, symptoms, functional capacity and quality of life related to health (HRQOL). Sixty patients will be randomized into the two groups: ERR starts the program during admission and continues at home immediately after discharge for a period of 3 months; CRR was started at home one month after discharge from hospital and continues for 3 months. Recruitment of patients and starting the RR program will occur in the first year. In the second year we will continue the intervention to those who have not completed the year. Follow-up will last until the completion of the year of all patients.

ELIGIBILITY:
Inclusion Criteria:

* Age> 40 years
* Diagnostic criteria of COPD GOLD II-IV confirmed by spirometry
* Having frequent re-admissions (≥ 2 times / year).
* Sign the informed consent.

Exclusion Criteria:

* Have completed a pulmonary rehabilitation program (including training) in the last 6 months.
* Respiratory and / or cardiac serious associated diseases.
* End-stage COPD (inability to perform exercises or treatment with morphine).
* Prognosis of <6 months.
* Living in a residence or not having a primary caregiver.
* Cognitive disorders that prevent active participation.
* Patients who are admired to other hospitalization rooms than Pneumology.
* Patients who do not belong to the area of health coverage of the Respiratory Rehabilitation home team

Ages: 41 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-06-09 (Actual); Study Completion 2017-06-09 (Actual)

PRIMARY OUTCOMES:
Exacerbations | 1 year
  Exacerbations with or without admission due to respiratory illness

SECONDARY OUTCOMES:
Dyspnea | 1 year
  dyspnea in activities of daily living measured by the area of the dyspnea in the original CRQ questionnaire
Functional capacity | 1 year
  Exercise capacity with the six minutes walk test
Quality of life related to health | 1 year
  Quality of life related to health from self-administered CAT and CRC questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Fátima E Morante, Nurse, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Servicio de Neumología Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

REFERENCES:
- [Derived] Guell-Rous MR, Morante-Velez F, Flotats-Farre G, Paz-Del Rio LD, Closa-Rusines C, Ouchi-Vernet D, Segura-Medina M, Bolibar-Ribas I. Timing of Pulmonary Rehabilitation in Readmitted Patients with Severe Chronic Obstructive Pulmonary Disease: A Randomized Clinical Trial. COPD. 2021 Feb;18(1):26-34. doi: 10.1080/15412555.2020.1856059. Epub 2020 Dec 7. PMID 33287581